CLINICAL TRIAL: NCT05057975
Title: Validation d'Une Solution Digitale intégrée (SUNrise®) d'Analyse Automatique Des Mouvements Mandibulaires Par Intelligence Artificielle Versus Polysomnographie Pour le Diagnostic du Syndrome d'Apnées Obstructives du Sommeil
Brief Title: Validation of an Integrated Digital Solution (SUNrise®) Versus Polysomnography for Obstructive Sleep Apnea Diagnosis
Acronym: SUNSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunrise (Industry)
Collaborators: ICUREsearch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-545
Record Dates: First submitted 2021-08-27; First posted 2021-09-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: polysomnography; obstructive sleep apnea; home sleep test; artificial intelligence; mandibular movement
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized, parrallel, open label, multicenter and national
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunrise (Experimental): Home Sleep Test, OSA diagnosis based on mandibular movements recording
  Interventions: Device: Sunrise
- PSG (Active Comparator): Polysomnography, OSA diagnosis based on local scoring by center
  Interventions: Device: polysomnography

INTERVENTIONS:
Device: Sunrise — Use of the Sunrise device for three nights to register mandibular movements that will be automatically analysed using artificial intelligence.
  Arms: Sunrise
Device: polysomnography — Reference protocol to diagnose OSA (in-lab or outpatient PSG)
  Arms: PSG

SUMMARY:
Validation of an integrated digital solution (SUNrise®) of mandibular movement automatic analysis by artificial intelligence versus polysomnography for obstructive sleep apnea diagnosis: a prospective, randomized, parallel-arm, open-label, multicenter, national, controlled study.

DETAILED DESCRIPTION:
The new Sunrise integrated digital solution is a disposable 3 gram sensor that sits on the chin for sleep disorders diagnosis. This device records mandibular movements, head movements and position during sleep. Data acquisition is done through a mobile application installed on the user smartphone. Data is then transferred automatically at the end of the test (overnight) to a cloud platform where it is automatically analyzed. The Health Care Professional (HCP) and the patient have access to sleep parameters and report.

The objective of this trial is to determine the place of the Sunrise device in the care pathway in France for patients suspected of having OSA. The assumption is that Sunrise is both non-inferior to the normal practice (i.e., the PSG) on sleepiness at 3 months post-diagnosis, and superior to the PSG (outpatient or in-lab) in terms of time between inclusion and diagnosis appointment and treatment initiation. By speeding up the treatment initiation, the hypothesis is that Sunrise is also superior to the PSG on sleepiness as well as quality of life and work productivity at 3 months post-inclusion. Another assumption is that Sunrise is non-inferior to the PSG on CPAP compliance at 3 months following treatment initiation.

The SUNSAS study will be launched in 19 centers (public and private) in France and will include 848 patients aged 18 to 80 years. Eligible patients will be included and randomized in 2 arms, i.e., the Sunrise arm and the PSG arm. An appointment to discuss the diagnosis and treatment options (for patients suffering from OSA) will be arranged after the procedure (PSG or Sunrise) is performed. On site follow-up visits will be then organized at 3 months post-inclusion and at 3 months post-diagnosis, and a phone call will be scheduled at 3 months post-treatment.

ELIGIBILITY:
Inclusion criteria:

* Man or woman aged between 18 to 80 years old
* Patient referred for a suspicion of OSA
* Patient having a smartphone and internet connection at home and able to use a mobile application
* Patient affiliated to the social security system

Main exclusion criteria:

* Patient with a previous sleep test performed within 5 years of inclusion
* Patient previously treated for OSA within 5 years of inclusion
* Patient suffering from severe chronic obstructive or restrictive pulmonary disease with or without oxygen at the discretion of the investigator
* Patient refusing to shave his beard that could prevent him to wear the device on the chin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Change in daily sleepiness | 3 months post-diagnosis
  To determine the non-inferiority of Sunrise vs PSG on sleepiness at 3 months post-diagnosis using the Epworth Sleepiness Scale (ESS) score.
  The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher the average sleep propensity in daily life.
Time to diagnosis | Up to 12 months
  To determine the superiority of Sunrise vs PSG in terms of time between inclusion and diagnosis appointment
Time to treatment | Up to 15 months
  To determine the superiority of Sunrise vs PSG in terms of time between inclusion and treatment initiation
Change in daily sleepiness | 3 months post inclusion
  To determine the superiority of Sunrise vs PSG on sleepiness at 3 months post-inclusion using ESS

SECONDARY OUTCOMES:
Change in quality of life | 3 months post inclusion visit
  To determine the superiority of Sunrise vs PSG on quality of life at 3 months post-inclusion using Short Form 36 (SF-36) SF-36 is a 0-100 scale score, a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in quality of life | 3 months post inclusion visit
  To determine the superiority of Sunrise vs PSG on quality of life at 3 months post-inclusion using Quebec Sleep Questionnaire (QSQ).
  QSQ utilizes 32 items to measure 5 domains: daytime sleepiness, diurnal symptoms, nocturnal symptoms, emotions, and social interactions.Item scores range from 1 to 7. Mean scores for each domain are calculated, and a total score is derived by calculating the mean of all items. Higher scores are associated with better better quality of life.
Change in work productivity | 3 months post-inclusion
  To determine the superiority of Sunrise vs PSG on work productivity at 3 months post-inclusion using WPAI:SHP
cost (€)/QALY | 3 months post-diagnosis
  cost (€)/QALY gained 3 months post-diagnosis
Net profit for the French social security | estimated at 3 years
  Estimation of the net profit for the French social security at 3 years
Comparison of CPAP compliance data | 3 month after treatment initiation
  To determine the non-inferiority of Sunrise vs PSG on CPAP compliance measured at 3 months post-treatment by comparing CPAP average usage in both groups
Comparison of Sunrise versus PSG diagnosis | Up to 12 months
  To confirm the diagnosis performance of Sunrise compared to PSG by comparing the obstructive respiratory disturbance index (ORDI) in both groups
Difference in the obstructive respiratory disturbance index (ORDI) | Up to 12 months
  To measure the variability of the ORDI by comparing the 3 obstructive respiratory disturbance index (ORDI) measures provided by the Sunrise device (used 3 nights)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Pr, Principal Investigator — CHU Grenoble Alpes
Locations (19):
- France (19):
  - CHU Angers, Angers
  - Hôpitaux Universitaires de Paris Seine Saint-Denis (HUPSSD, AP-HP),, Bobigny
  - Nouvelle clinique Bel-Air, Bordeaux
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - AP-HP Hôpital Henri Mondor, Créteil
  - Chu Grenoble Alpes,, Grenoble
  - CHRU Lille - Hôpital Roger Salengro, Lille
  - Hôpital privé la Louvière, Lille
  - CHU Lyon - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Européen Marseille, Marseille
  - CHU Montpellier - Hôpital Gui-de-Chauliac, Montpellier
  - CHRU de Nancy - Hôpital d'Adultes de Brabois, Nancy
  - AP-HP Pitié Salpêtrière, Paris
  - AP-HP Hôpital Bichat-Claude Bernard, Paris
  - AP-HP CUP Hôpital Hôtel Dieu, Paris
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - Polyclinique Saint-Laurent, Rennes
  - Centre du Sommeil de Grenoble, Saint-Martin-d'Hères
  - CHU de Toulouse - Hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: No